CLINICAL TRIAL: NCT05474950
Title: Efficacy and Safety of the Treatment of Minocycline for Cystoid Macular Edema
Brief Title: Minocycline Treatment for Cystoid Macular Edema
Acronym: MINOCME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Dan Liang, PhD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MINOCME
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Minocycline; Cystoid Macular Edema
MeSH Terms: conditions — cyclopia sequence; Macular Edema | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- minocycline (Experimental)
  Interventions: Drug: minocycline

INTERVENTIONS:
Drug: minocycline — minocycline capsule (100mg) per day orally

SUMMARY:
Cystoid macular edema (CME) is one of sight-threatening, immune-related ocular diseases. The efficacy of current treatments for CME (anti-VEGF, glucocorticoids and other agents) are limiting. Minocycline, acting as a broad-spectrum antibiotic, is among tetracycline family and recently, its immunomodulatory and anti-apoptosis function has been replied to several immune diseases and degenerative diseases. This study aims to explore the efficacy and safety of minocycline for CME.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with CME.
* Participant aged from 18-60 years old.
* Participant that signed the informed consent document and is able to complete the following visits.

Exclusion Criteria:

* Participant is allergy to minocycline or tetracyclines.
* Participant has no contraindications of minocycline or tetracyclines.
* Participant has an abnormal function of liver, heart, kidney and thyroid.
* Female that is pregnant, breast-feeding or planning to become pregnant.
* Participant that is currently using other medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of cystoid macular edema | At 6 months
  Change of CME measured by Optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Change of best corrected visual acuity (BCVA) | At 6 months
  Change of BCVA measured by the Early Treatment Diabetic Retinopathy Study
Change of macular sensitivity | At 6 months
  Change of BCVA measured by Macular Integrity Assessment (MAIA)
Change of retinal vascular leakage | At 6 months
  Change of retinal vascular leakage measured by Fundus fluorescein angiography (FFA) or indocyanine green angiography (ICGA)
Change of macular vessel | At 6 months
  Change of macular vessel measured by optical coherence tomography angiography (OCTA)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792